CLINICAL TRIAL: NCT04695704
Title: Double-blind Randomized Clinical Trial, Placebo-controlled to Assess the Efficacy of Montelukast in Mild-moderate Respiratory Symptoms in Patients With Long-COVID-19: E-SPERANZA COVID-19 PROJECT
Brief Title: Efficacy of Montelukast in Mild-moderate Respiratory Symptoms in Patients With Long-COVID-19:
Acronym: E-SPERANZA
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The incidence of respiratory Long COVID has decreased in the new waves, thus made impossible to achieve the required study sample.
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Collaborators: Institut Català de la Salut (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 4R21/006
Record Dates: First submitted 2021-01-04; First posted 2021-01-05 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Covid19; SARS (Disease)
Keywords: SARS-CoV-2; Montelukast; Leukotriene Antagonists; Primary Health Care; Clinical Trial; Quality of Life; Long Term Covid
MeSH Terms: conditions — COVID-19; Severe Acute Respiratory Syndrome; Disease | interventions — montelukast

STUDY DESIGN:
Intervention Model Description: Double-blind randomized placebo-controlled clinical trial,.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple (Participant, Care Provider, Investigator and Outcomes Assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Montelukast (Experimental): 10mg oral montelukast once daily for 28 days.
  Interventions: Drug: Montelukast
- Placebo (Placebo Comparator): oral placebo once daily for 28 days.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Montelukast — 10 mg oral montelukast once daily for 28 days
  Other Names: antileukotriene
  Arms: Montelukast
Other: placebo — 10 mg oral placebo once daily for 28 days
  Arms: Placebo

SUMMARY:
Recently, a new clinical presentation called "long covid" has been reported, for patients with symptoms lasting for more than 4 weeks from the onset of the disease. Typically, the symptoms comprise dyspnea, cough, headache, arthralgia, fever, abdominal pain, asthenia and skin manifestations This project aims to evaluate the efficacy of Montelukast in improving the quality of life associated with respiratory symptoms in patients with persistent COVID-19 symptoms. The main objective is to compare the efficacy of low-dose Montelukast versus placebo to improve respiratory symptoms in patients with persistent COVID-19 symptoms.

DETAILED DESCRIPTION:
In December 2019, the first case of a new coronavirus causing pneumonia was described in Wuhan (China), designated as SARS-CoV-2 by the World Health Organization.

From the start of the SARS-CoV-2 alert until May 21st, 2020, 250,287 cases of coronavirus disease (COVID-19) were reported in Spain. The importance of the COVID-19 pandemic with its high humanitarian and economic cost, urgently requires effective therapies to reduce the severity, complications and mortality associated with this infection.

As the number of cases of COVID-19 increases, so does information regarding the management and evolution of the disease. More recently, a new clinical presentation called "long COVID-19" has been reported, for patients with symptoms lasting for more than 4 weeks from the onset of the disease. Typically, the symptoms comprise dyspnea, cough, headache, arthralgia, fever, abdominal pain, asthenia and skin manifestations.

The inflammatory process produced at the pulmonary and extra pulmonary level, and the immune response triggered have been identified as important mechanisms in the pathophysiology of COVID-19.

Coronavirus infection activates the cytokine cascade at the immune level, in which leukotriene are possibly involved in the development of respiratory symptoms in patients with persistent symptoms after infection by SARS-CoV-2.

Leukotriene antagonists (LTRAs) have a bronchodilator action and inhibit inflammation of the airways, resulting in a significant improvement in asthma symptoms and allergic rhinitis. In asthma, they improve respiratory function, inhalation rate of inhaled β2 agonist, airway inflammation, airway hyper responsiveness, inhaled corticosteroid dosage, and reduce exacerbations.

Regarding the treatment of acute SARS-CoV-2 infection, to date, the available evidence is limited; there are few conclusive clinical trials that allow recommendations based on scientific evidence.

To date, no treatment has been evaluated in long COVID-19. The hypothesis of using Montelukast would be based on the pathophysiological response of the disease mediated by the immune system against the SARS-CoV-2 infection.

Montelukast blocks the action of substances such as leukotriene C4, D4 and E4 by binding to the CysLT1 receptor in the lungs and bronchi. This reduces the bronchoconstriction caused by leukotriene and results in less inflammation.

Montelukast effectively attenuated both lung inflammation induced by Lipopolysaccharides in a mouse model with Acute Respiratory Distress Syndrome, as in human neutrophils.

Individuals affected by long COVID-19 have self-organized to gain visibility. They have made a self-completed form to describe the characteristics of the disease. The "Persistent COVID19" network in Catalonia currently gathers more than 3000 people.

From the contact with the "Persistent COVID19 association" in Catalonia, and in search of a response to this symptomatology, which can be very disabling, a pilot study was carried out in patients with persistent COVID-19 symptoms with off-label use of Montelukast.

Empirical treatment with Montelukast at a dose of 10 mg / day for 14 days was started in 13 patients with long COVID-19, some with symptoms of more than a month of evolution since the beginning of the COVID-19 clinic. The patients were followed up to evaluate the improvement of the symptoms with a numerical scale from 0 to 100 and COPD Assessment Test Scale (CAT), 3 weeks after starting treatment.

An improvement in symptoms was observed a few days after treatment and a good evolution of the sensation of dyspnea, chest pain, symptoms of discomfort, dry cough, and nasal symptoms. Likewise, the incorporation of the patients to their work activity during that period was observed. To date, the improvement continues to exist, without evidence of clinical deterioration.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 to 80 years old with SARS-CoV-2 infection (positive CRP <10 days from the onset of symptoms) treated in Primary Health Care.
* Persistent respiratory symptoms (more than 1 and <12 months of evolution)
* Mild-moderate dyspnea: score at the beginning of the study according to the modified Medical Research Council (mMRC) scale from 0 to 3
* The patient must be competent to complement the follow-up evaluations.
* The patient agrees to participate in the study and take assigned medication during the 4 weeks.
* Sign the informed consent

Exclusion Criteria:

* Severity criteria: fever> 38ºC, or O2 saturation <93%.
* Patients with SARS-Cov-2 pneumonia in the acute / subacute phase.
* Patients who have required hospital admission for SARS-Cov-2.
* Chronic Obstructive Pulmonary Disease (COPD), asthma, bronchiectasis, pulmonary fibrosis, obstructive sleep apnea syndrome (OSAS), chronic respiratory failure from any cause, home oxygen therapy.
* Use of montelukast or zafirlukast ≤ 30 days prior to inclusion
* Use of any dose of systemic corticosteroids ≤ 30 days prior to inclusion
* Use of gemfibrocil.
* Hypersensitivity to montelukast or to any of the excipients included (e.g. lactose.
* Any condition (including the inability to swallow pills) that, in the opinion of the researcher, would prevent the completion of taking the medication.
* Active malignancy, current or recent chemotherapy treatment (<6 months).
* Medical history of infection by the Human Immunodeficiency Virus (HIV) or any serious immunocompromised state.
* Pregnancy, planning to get pregnant or patients of childbearing age not undergoing birth control methods.
* Breastfeeding mother.
* Any other condition for which, in the opinion of the principal investigator, it is considered that the subject does not fit the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2021-08-11 (Actual); Primary Completion 2023-07-24 (Actual); Study Completion 2023-08-28 (Actual)

PRIMARY OUTCOMES:
COP Assessment Test Scale (CAT) | 7, 14, 21 and 28 days
  Quality of life of respiratory symptoms according to COPD Assessment Test (CAT The COPD Assessment Test (CAT) is a questionnaire for people with COPD, designed to measure the impact of COPD on a person's life, and how this changes over time.Quality of life of respiratory symptoms according to COPD Assessment Test (CAT). This is a validated self-administered scale to quantify and monitor the impact of COPD on well-being and daily life. It consists of 8 items (from 0 to 5 points), and a total score of 0-40 (0-9 mild, 10-20 moderate, 21-30 severe and 31-40 very severe), being higher scores worse outcome. A difference of 2 or more points in health status is considered clinically significant.

SECONDARY OUTCOMES:
1min sit-to-stand test | 14 and 28 days
  Exercise capacity: number of repetitions performed in the 1min sit-to-stand test
O2 desaturation | 14 and 28 days
  O2 desaturation ≥ 4% with effort (1min sit-to-stand test)
Visual Analogical Scale (VAS) | 7, 14, 21 and 28 days
  Symptoms evaluated using numeric Visual Analogical Scale (VAS): asthenia, headache, ageusia, anosmia, and rhinitis . It is numbered from 0-10, where 0 is the absence and 10 the greatest intensity, meaning higher scores worse outcome. The patient selects the number that best evaluates the intensity of the symptom.
All-cause mortality | 7, 14, 21 and 28 days
  Mortality from any cause during the study
Number of visits to primary care | 28 days
  Number of visits of any kind to primary health care settings (phone visit or face to face visit) during the study period.
Number of visits to the emergency room | 28 days
  Number of visits to emergency room form primary health o hospital settings during the study period.
Number of hospital admissions. | 28 days
  Number of hospital admissions during the study period.
Medication side effects | 7, 14, 21 and 28 days
  Number and type of adverse reactions during the study period related to medication.
Days of sick leave | 28 days
  Number of days of incapacity for work (sick leave) during the study period.
Factors of inflamatory and prothrombotic processes: D-Dimer, N-terminal prohormone of brain natriuretic peptide (NT Pro-BNP), C-reactive protenin and Antinuclear antibodies (ANA) | 0 and 28 days
  To analyze wether the factors of inflamatory and prothrombotic processes (D-Dimer, Pro-BNP, C-reactive protein, and ANA) at the begining of the study are response predictors to the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jesus Almeda Ortega, PhD, Study Chair — Institut Català de la Salut; Sara Bonet Monne, PhD, Study Chair — Institut Català de la Salut; Betlem Salvador Gonzalez, PhD, Study Chair — Institut Català de la Salut; Francisco Mera Cordero, MD, Principal Investigator — Institut Català de la Salut
Locations (8):
- Spain (8):
  - Primaty health Center Corbera, Corbera de Llobregat, Barcelona
  - Primary Health Center Jaume Soler, Cornellà de Llobregat, Barcelona
  - Primary Health Center 17 Setember, el Prat de Llobregat, Barcelona
  - Primary Health Center Camps Blancs, Sant Boi de Llobregat, Barcelona
  - Primary Health Center Molí Nou, Sant Boi de Llobregat, Barcelona
  - Primary Health Center Vinyets, Sant Boi de Llobregat, Barcelona
  - Primary Health Center ElPla, Sant Feliu de Llobregat, Barcelona
  - Primary Health Center Raval nord, Barcelona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mera-Cordero F, Bonet-Monne S, Almeda-Ortega J, Garcia-Sangenis A, Cunillera-Puertolas O, Contreras-Martos S, Alvarez-Munoz G, Monfa R, Balanzo-Joue M, Morros R, Salvador-Gonzalez B. Double-blind placebo-controlled randomized clinical trial to assess the efficacy of montelukast in mild to moderate respiratory symptoms of patients with long COVID: E-SPERANZA COVID Project study protocol. Trials. 2022 Jan 6;23(1):19. doi: 10.1186/s13063-021-05951-w. PMID 34991703